CLINICAL TRIAL: NCT05969899
Title: Prospective and Exploratory Study of Liposomal Irinotecan Based FOLFIRI Combined With Bevacizumab in First-line Treatment of Advanced Colorectal Cancer
Brief Title: Liposomal Irinotecan Based FOLFIRI With Bevacizumab in First-line Treatment of Advanced Colorectal Cancer
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, LI XIN-XIANG, Head of the second ward of colorectal Surgery, Fudan University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MA-CRC-II-008
Record Dates: First submitted 2023-07-19; First posted 2023-08-01 (Actual); Last update posted 2024-11-21 (Actual); Status verified 2024-11

CONDITIONS: Colorectal Cancer
Keywords: irinotecan liposome; FOLFIRI
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- FOLFIRI+BEV (Other)
  Interventions: Drug: FOLFIRI+Bevacizumab

INTERVENTIONS:
Drug: FOLFIRI+Bevacizumab — irinotecan liposome 60 mg/m2, iv, for at least 90 minutes LV 400 mg/m2, iv, for at least 2 hours FU 400 mg/m2, iv, followed by FU 2400 mg/m2, iv for at least 46 hours bevacizumab 5mg/kg IV. The above scenario is repeated every two weeks. Patients were treated until disease progression, toxic intolerance, initiation of a new antitumor therapy, withdrawal of knowledge, or investigator judgment that subjects should withdraw from study therapy.

SUMMARY:
The goal of this prospective clinical trial is to evaluate efficacy and safety of irinotecan liposomes for first-line treatment of advanced colorectal cancer. The primary endpoint is Objective response rate (ORR) per RECIST 1.1. The secondary endpoints are overall survival (OS), progression-free survival (PFS), disease control rate (DCR) and safety based on NCI-CTCAE 5.0

ELIGIBILITY:
Inclusion Criteria:

1. Provide written informed consent to participate in the study voluntarily.
2. Male or female aged 18-75.
3. Metastatic colorectal adenocarcinoma confirmed by histology or cytology.
4. Have not received systematic anti-tumor therapy before; Patients who have received neoadjuvant/adjuvant therapy may be screened from the time of last chemotherapy to recurrence or progression more than 6 months.
5. RAS/BRAF mutation status and UGT1A1*28/*6 gene polymorphism typing should be determined before enrollment.
6. The ECOG PS score is 0 or 1.
7. Life expectancy is at least 3 months.
8. According to RECIST 1.1, the investigators evaluated that there were measurable lesions at baseline (according to RECIST 1.1), which could be measured if they had not received local treatment such as radiotherapy (lesions located within the area of previous radiotherapy could also be selected as target lesions if progression was confirmed).
9. The function of vital organs meets the following requirements (no blood component, cell growth factor correction therapy drugs are allowed within 14 days before the first use of the study drug);

   1. Absolute neutrophil count (ANC) ≥1.5×109/L
   2. Platelet ≥100×109/L;
   3. Hemoglobin ≥9g/dL;
   4. Serum albumin ≥2.5g/dL;
   5. Total bilirubin ≤1.5 × ULN; ALT and AST≤2.5 × ULN, if there is liver metastasis, ALT and AST≤5 × ULN;
   6. Serum creatinine ≤1.5 × ULN or creatinine clearance > 60 mL/min (Cockcroft-Gault);
   7. Activated partial thromboplastin time (APTT) and International Normalized ratio (INR) ≤1.5 × ULN (for stable dose anticoagulant therapy such as low molecular weight heparin or warfarin and INR within the intended therapeutic range of anticoagulants can be screened)
10. Fertile female subjects are required to have a negative serum pregnancy test within 72 hours before the first dosing, are not breastfeeding, and use effective contraception (such as Iuds, contraceptives, or condoms) during the trial period and for at least 6 months after the last dosing of the study drug; Male subjects whose partner is a fertile woman should be surgically sterilized or agree to use effective contraception during the trial period and within 3 months after the last dose of the study drug. Sperm donation is not allowed during the study period;

Exclusion Criteria:

1. Local radiotherapy was received within 4 weeks prior to the first administration of the study drug, and adverse events due to radiotherapy have not returned to baseline levels. Participants who received palliative radiotherapy for peripheral sites (such as bone metastases) before 4 weeks may be admitted to the study, but must have recovered from any acute adverse effects;
2. Known active central nervous system (CNS) metastases and/or cancerous meningitis. Participants who have previously received BMS may participate in treatment provided they have stable BMS and have not been treated with steroids for BMS for at least 28 days prior to study start. This exception does not include cancerous meningitis, as patients with cancerous meningitis are excluded regardless of clinical stability;
3. Major surgery, open biopsy, or severe trauma occurred 28 days before the first medication;
4. Previous history of allergy to fluorouracil or irinotecan;
5. Have high blood pressure that is not well controlled by antihypertensive medication (systolic blood pressure ≥140 mmHg or diastolic blood pressure ≥90 mmHg)
6. Subjects have poorly controlled cardiovascular clinical symptoms or diseases, including but not limited to:

(1) NYHA grade II or above heart failure; (2) unstable angina pectoris; (3) myocardial infarction within 1 year; (4) Clinically significant supraventricular or ventricular arrhythmias that remain poorly controlled without or after clinical intervention.

7. Clinically significant bleeding symptoms or definite bleeding tendency, such as gastrointestinal bleeding, hemorrhagic ulcer or vasculitis, have occurred within 3 months before the first medication.

8. Arteriovenous thrombosis events occurring within 6 months before the first medication, such as cerebrovascular accidents (including temporary ischemic attack, cerebral hemorrhage, and cerebral infarction), deep vein thrombosis and pulmonary embolism, etc. Shallow vein thrombosis can be included after being determined by the researcher.

9. There is another malignant tumor that is progressing or in need of aggressive treatment, except for non-melanoma skin cancer and cervical cancer in situ for which potential treatment has been performed.

10. In the investigator's judgment, the subject has other factors that may lead to the forced termination of the study, such as other serious medical conditions (including mental illness) requiring co-treatment, serious abnormalities in laboratory test values, and family or social factors that may affect the subject's safety or the circumstances in which the trial data are collected.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-07-10 (Actual); Primary Completion 2025-07-10 (Estimated); Study Completion 2027-02-10 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate（ORR） | up to 2.5 years
  The proportion of participants in the analyzed population who developed complete (CR) or partial response (PR) according to RECIST 1.1 criteria

SECONDARY OUTCOMES:
Overall Survival（OS） | up to 2.5 years
  From the time of patient admission to the time of subject's death, at the end of the study, if the subject is still alive, the last known date of subject's survival is the deletion date
Progression Free Survival（PFS） | up to 2.5 years
  Time from patient admission to first radiographic disease progression (RECIST 1.1 criteria) or death (whichever occurs first)
Disease Control Rate（DCR） | up to 2.5 years
  The proportion of subjects in the analyzed population who achieved CR, PR, or stable disease (SD) according to RECIST 1.1 criteria

CONTACTS AND LOCATIONS:
Overall Officials: Xinxiang li, PhD, Principal Investigator — Affiliated Cancer Hospital of Fudan University
Locations (1):
- Affiliated Cancer Hospital of Fudan University, Shanghai, Pudong, China

IPD SHARING:
Plan to Share IPD: No